CLINICAL TRIAL: NCT03441776
Title: Towards Comparative Effectiveness in Military Vestibular Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Collaborators: Evans Army Community Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHC-A-18-006
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Vestibular Problem; Traumatic Brain Injury
Keywords: TBI; Rehabilitation; Vestibular; Dizziness
MeSH Terms: conditions — Vestibular Diseases; Brain Injuries, Traumatic; Dizziness

STUDY DESIGN:
Intervention Model Description: This is a single site, randomized, open label, pilot study to test the environment, resources and tools required to perform a comparative effectiveness trial assessing two different standard of care vestibular rehabilitation approaches.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Randomized GVRT (Other): Randomized Generalized Vestibular Rehabilitation Treatment (8 treatments) as part of standard of care (not research visits)
  Interventions: Other: Generalized Vestibular Rehabilitation Treatment
- Randomized IVRT (Other): Randomized Individualized Vestibular Rehabilitation Treatment (3 treatments) as part of standard of care (not research visits)
  Interventions: Other: Individualized Vestibular Rehabilitation Treatment

INTERVENTIONS:
Other: Generalized Vestibular Rehabilitation Treatment — These treatment visits are available twice a week and each visit lasts 45 minutes. Individuals receiving GVRT are allowed to choose the frequency at which they want to attend and the program is designed for each subject to complete 8 visits within a period between 4 and 8 weeks. The ideal number of patients receiving treatment at each class is from 3 to 6 but the system has capacity for a maximum of 8. GVRT is a standard of care treatment option and is not considered research.
  Other Names: GVRT
  Arms: Randomized GVRT
Other: Individualized Vestibular Rehabilitation Treatment — Individuals receiving IVRT are scheduled depending on their individual needs and PT availability. These visits require one-on-one time with a PT. Individuals are commonly seen by the PT 3 times at two week intervals. These visits last 30 minutes and include PT evaluation designed to instruct patients on exercises for them to perform on their own. IVRT is a standard of care treatment option and is not considered research.
  Other Names: IVRT
  Arms: Randomized IVRT

SUMMARY:
To prospectively evaluate the tools, environment and resources to compare the effectiveness of two different standard of care vestibular rehabilitation approaches in a military cohort with post-concussive vestibular symptoms.

DETAILED DESCRIPTION:
Aim 1. To prospectively evaluate the reliability of a series of diagnostic and outcome assessment tools in a military cohort with post-concussive vestibular symptoms; these to include the Dizziness Handicap Inventory (DHI), Activities-Specific Balance Confidence Scale (ABC), the Computerized Dynamic Posturography (CDP) and the Neuro-Otologic Test System (NOTC).

Hypothesis 1. Active military personnel consist of physically high functioning individuals in whom standard diagnostic and outcome assessment tools may fail to target variations in performance. The investigators believe that active military personnel score different than general populations in standard diagnostic and outcome assessment tools.

Endpoint 1. The investigators will compare the DHI, ABC, CDP and NOTC results obtained in this study with historical data from the studies supporting the validation of each of the individual assessment tools.

Aim 2. To assess the concept of 'clinically meaningful change' as it relates to dizziness specific to a military cohort with post-concussive vestibular symptoms.

Hypothesis 2. Because of the differences in physical characteristics and performance demands between active duty military personnel and the general population, it is difficult to define if changes in diagnostic and outcome assessment evaluations in the military population reflect worsening or progression of symptoms at the same rate and magnitude observed in the general population.

Endpoint 2. The investigators will establish a comparison among study test results (DHI, ABC, CDP and NOTC) and compare these to clinical measures of response to treatment (Neurobehavioral Symptom Inventory - vestibular domain and Patients' Global Impression of Change Scale) to identify the rate and magnitude of change in the military cohort.

Aim 3. To compare scoring differences between subjects receiving individualized vestibular rehabilitation treatment (IVRT) and subjects receiving generalized vestibular rehabilitation treatment (GVRT), and to calculate the magnitude of change or the lack of it to determine the sample size for a subsequent comparative effectiveness trial.

Hypothesis 3. The combination of tests used in this study has not been used before; therefore, no data is available to calculate the sample size needed to determine comparative effectiveness between GVRT vs IVRT using DHI, ABC, CDP and NOTC.

Endpoint 3. The investigators will compare DHI, ABC, CDP and NOTC measurement results between treatment groups to estimate normal variation.

Aim 4. To refine methods, procedures, and information parameters for a comparative effectiveness trial assessing individualized vs. generalized vestibular rehabilitation therapy.

Endpoint 4. The investigators will evaluate and compare different elements inherent to the trial such as mechanisms of subject identification, evaluation times and tolerance, information tracking, etc. along with data obtained through the Patient Satisfaction Survey (PSS).

ELIGIBILITY:
Inclusion Criteria:

* Active Duty Service Member
* Referral to Warrior Recovery Center
* Need of treatment for gaze stabilization, static standing, balance, dynamic standing balance, gait, motion sensitivity, modified center of gravity, and/or work-related functional task training; determined by physical therapist
* Dizziness as identified by a score of 16 - 64 on DHI
* Personal history of Mild-Traumatic TBI occurring between 4 weeks and 5 years from the Pre-Treatment PT Evaluation Visit
* Fluency in English

Exclusion Criteria:

* Participation in a concurrent interventional trial
* History of Severe TBI
* Inability to participate in treatment visits or any of the research activities
* Any vestibular dysfunction that cannot be treated with a generalized treatment plan (e.g. benign paroxysmal positional vertigo, acute vestibular infection) as defined by PT discretion
* Any unstable and/or chronic medical or psychiatric condition that could confound the results of the study and/or place the participant at risk

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change in Dizziness Handicap Inventory (DHI) score | Baseline and 2 weeks after final treatment visit
  Self reported perception of handicap related to dizziness. 25 questions. Each item is scored 0 - 4 (0 = no, 2 = sometimes, 4 = always), yielding a total score between 0 (no perceived disability) and 100 (maximum perceived disability). Subscales related to certain questions are describes as physical, emotional and functional disabilities.

SECONDARY OUTCOMES:
Change in Activities-specific Balance Confidence (ABC) Scale | Baseline and 2 weeks after final treatment visit
  Self reported level of confidence of not losing balance or becoming unsteady during specific activities. Participants rate their perceived confidence on a 0-100% scale (0% = no confidence, 100% = completely confident). Total score is averaged percentage of 16 questions.
Change in Equilibrium Score on Sensory Organization Test (SOT) | Baseline and 2 weeks after final treatment visit
  Equilibrium score quantifies postural stability during each of 3 trials of 6 sensory conditions obtained via Computerized Dynamic Posturography (CDP). Equilibrium is scored between 0 and 100 (0 = worst, 100 best).
Change in Composite Equilibrium Score on Sensory Organization Test (SOT) | Baseline and 2 weeks after final treatment visit
  Composite Equilibrium Score is averaged from the six SOT Equilibrium Scores. Equilibrium score quantifies postural stability during each of 3 trials of 6 sensory conditions obtained via Computerized Dynamic Posturography (CDP). Equilibrium is scored between 0 and 100 (0 = worst, 100 best).
Change in Equilibrium Score on Horizontal Head-Shake Sensory Organization Test (HS-SOT) | Baseline and 2 weeks after final treatment visit
  Equilibrium score quantifies postural stability with horizontal head movement during each of 3-4 trials of 2 sensory conditions obtained via Computerized Dynamic Posturography (CDP). Equilibrium is scored between 0 and 100 (0 = worst, 100 best).
Change in Equilibrium Score Ratio (SOT and Horizontal HS-SOT) | Baseline and 2 weeks after final treatment visit
  Equilibrium Score Ratio compares the average Equilibrium Score between the SOT and HS-SOT relating to the same sensory conditions. Equilibrium score quantifies postural stability during each of 3-4 trials of 2 sensory conditions obtained via Computerized Dynamic Posturography (CDP). Equilibrium is scored between 0 and 100 (0 = worst, 100 best).
Change in logMAR (Visual Acuity) during horizontal head movement (Dynamic Visual Acuity) | Baseline and 2 weeks after final treatment visit
  logMAR is given for positive and negative responses during left movement and right movement. logMAR is a unit describing the apparent size of an image based on a ratio of its absolute size to distance from the eye.
Change in logMAR (Visual Acuity) during vertical head movement (Dynamic Visual Acuity) | Baseline and 2 weeks after final treatment visit
  logMAR is given for positive and negative responses during up movement and down movement. logMAR is a unit describing the apparent size of an image based on a ratio of its absolute size to distance from the eye.
Change in Neuro-Otologic Testing | Baseline and 2 weeks after final treatment visit
  Gaze Horizontal, Random Saccades Horizontal and Vertical, Smooth Pursuit Horizontal 0.1Hz and 0.75Hz, Smooth Pursuit Vertical 0.1Hz and 0.75Hz, Predictive Saccades Horizontal, Antisaccades, OKN Trap 20deg/sec and 60deg/sec, Visual Reaction Time, Saccade and Reaction Time, Auditory Reaction Time, Chair Rotation Sinusoidal 0.02Hz, 0.08Hz and 0.64Hz, Visual Enhancement, Visual Suppression, Step Test, Subjective Visual Vertical, crHIT

CONTACTS AND LOCATIONS:
Locations (1):
- Warrior Recovery Center, Evans Army Community Hospital, Fort Carson, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT03441776/ICF_000.pdf